CLINICAL TRIAL: NCT06626763
Title: Comparison of Oxygen Saturation Measurements Using Different Glove Colors in Children: A Preventive Method for Infection?
Brief Title: Comparison of Oxygen Saturation Measurements Using Different Glove Colors in Children
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ELİZ GECTAN, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 1753
Record Dates: First submitted 2024-09-29; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Infection; Oxygen Saturation; Children
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Children will be measured 5 times using a pulse oximeter. The measurements will be performed consecutively without any interval between them. The first measurement will be performed without using any gloves on the patient's finger, the second measurement will be performed using transparent gloves, the third measurement will be performed using white gloves, the fourth measurement will be performed using black gloves, and the fifth measurement will be performed using blue gloves.

SUMMARY:
The aim of this study was to determine the effect of different colored gloves on oxygen saturation in pediatric patients whose oxygen saturation was measured by pulse oximetry in pediatric emergency department. The population of the study, which is planned as a prospective cohort study, will consist of children between the ages of 3-18 years who underwent oxygen saturation measurements in the pediatric emergency clinic of İzmir Bakırçay University Cigli and Training and Research Hospital between October 2024 and October 2025.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of different colored gloves on oxygen saturation in pediatric patients who underwent oxygen saturation measurement by pulse oximetry in pediatric emergency department. The population of the study, which is planned as a prospective cohort study, will consist of children aged 3-18 years who underwent oxygen saturation measurements in the pediatric emergency clinic of İzmir Bakırçay University Çiğli and Training and Research Hospital between October 2024 and October 2025. The sample of the study will consist of children who meet the inclusion criteria on the specified dates and whose parents/legal guardians agree to participate in the study. Descriptive Characteristics Form and Oxygen Saturation Measurement Value Record Form will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3-18,
* The parent/legal guardian or the child himself/herself agrees to participate in the study,
* Arterial blood gas measurement was performed,

Exclusion Criteria:

* The finger has a skin condition,
* Having nail polish on your fingernails,
* Having a severed finger,

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children between the ages of 3-18
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2025-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Measuring the arterial blood gas SpO2 saturation | Procedure
  Finger SpO2 measurements will be initiated as soon as the blood gas measurement process starts. Pulse oximetry measurements and intra-arterial blood gas measurements will be performed
without gloves measuring the SpO2 saturation | While the patient was not wearing gloves, the pulse oximeter light source was placed on the outer surface of the finger. SpO2 was read after waiting an average of 30 seconds.
SpO2 saturation measurement with transparent colored glove | While the patient was wearing a transparent glove, the pulse oximeter light source was placed on the outer surface of the finger. SpO2 was read after waiting an average of 30 seconds.
SpO2 saturation measurement with white colored glove | While the patient was wearing a white glove, the pulse oximeter light source was placed on the outer surface of the finger. SpO2 was read after waiting an average of 30 seconds.
SpO2 saturation measurement with black colored glove | While the patient was wearing a black glove, the pulse oximeter light source was placed on the outer surface of the finger. SpO2 was read after waiting an average of 30 seconds.
SpO2 saturation measurement with blue colored glove | While the patient was wearing a blue glove, the pulse oximeter light source was placed on the outer surface of the finger. SpO2 was read after waiting an average of 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmirKCU, Izmir, Turkey (Türkiye)